CLINICAL TRIAL: NCT03020004
Title: A Phase 2,Multicenter,Open-Label Study to Investigate the Efficacy, Safety and Pharmacokinetics of Ritonavir-boosted Danoprevir in Combination With Peg-IFN and RBV in Treatment-Naive Non-Cirrhotic Patients Who Have Chronic Hepatitis GT1
Brief Title: Efficacy and Safety of Danoprevir/r + PR 12-week Triple Therapy in Treatment-Naive, Non-Cirrhotic, G1 CHC China II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Ascletis Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Ascletis Pharma Inc (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ASC08201502
Record Dates: First submitted 2017-01-05; First posted 2017-01-13 (Estimated); Results first posted 2018-02-07 (Actual); Last update posted 2018-07-26 (Actual); Status verified 2017-01

CONDITIONS: Chronic Hepatitis C
Keywords: Danoprevir; SVR12; Chinese HCV G1; non-cirrhotic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — danoprevir; Ritonavir; peginterferon alfa-2a; Ribavirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Danoprevir,Ritonavir, Peg-IFN,RBV (Experimental): Participants will receive a combination of Ritonavir-boosted Danoprevir 100mg/100mg BID, subcutaneous injection of weekly peginterferon alfa-2a at 180 mcg and oral Ribavirin (RBV)1000/1200 mg/day (bodyweight<75/≥75 kg) for 12 weeks.
  Interventions: Drug: Danoprevir; Drug: Ritonavir; Drug: peginterferon alfa-2a; Drug: Ribavirin (RBV)

INTERVENTIONS:
Drug: Danoprevir — Danoprevir (DNV) 100mg tablet administered orally twice daily
  Other Names: ASC08
Drug: Ritonavir — Ritonavir 100mg tablet administered orally twice daily
Drug: peginterferon alfa-2a — PegIFN subcutaneous injection at 180 mcg weekly
  Other Names: PegIFN
Drug: Ribavirin (RBV) — Ribavirin (RBV)1000/1200 mg/day (bodyweight<75/≥75 kg)
  Other Names: Ribasphere®

SUMMARY:
The purpose of this study is to evaluate the Efficacy, Safety and Pharmacokinetics of Ritonavir-boosted Danoprevir (ASC08) in Combination with Peg-IFN and RBV in Treatment-Naive Non-Cirrhotic Patients Who Have Chronic Hepatitis Genotype 1.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide written informed consent
* Chronic HCV infection (≥ 6 months) ;
* Positive HCV antibody
* Serum HCV RNA of ≥ 1 × 104 IU/mL
* Hepatitis C virus GT1
* Never received prior-treatment for HCV with interferon, RBV, or other direct-acting or host-targeting antivirals for HCV
* The liver biopsy methods in the protocol (non-cirrhosis is defined as: Metavir score ˂ 4), or as determined by Fibroscan defined as: ˂ 14.6 kPa. Patients who have not obtained a liver biopsy or Fibroscan in the last 1 years will have a study related Fibroscan performed in order to confirm the diagnosis
* Others as specified in the detailed protocol

Exclusion Criteria:

* Patients with Fibroscan detection value > 12.9 kPa, or histologic examination for liver cirrhosis patients
* Presence or history of non-hepatitis C chronic liver disease, including but not limited to, autoimmune hepatitis, α-1-antitrypsin deficiency, C282Y homozygous hemochromatosis, Wilson's disease, drug- or toxin-induced liver disease, alcohol-related liver disease, primary biliary cirrhosis, sclerosing cholangitis, and porphyria cutanea tarda causing liver pathology or requiring phlebotomy
* Patients with a history of liver cell cancer, screening before or screening suspected hepatocellular carcinoma (HCC) patients, or imaging studies found suspicious nodules, or AFP > 50 ng/mL
* Positive hepatitis A antibody，positive hepatitis B surface antigen，syphilis antibody or HIV antibody at screening
* Others as specified in the detailed protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2016-01; Primary Completion 2016-11 (Actual); Study Completion 2017-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Huoling Tang, PhD, Study Director — Ascletis Pharmaceuticals Co., Ltd.

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Danoprevir,Ritonavir, Peg-IFN,RBV
Started | 70
Completed | 69
Not Completed | 1

BASELINE CHARACTERISTICS:
Arm/Group | Danoprevir,Ritonavir, Peg-IFN,RBV
Number analyzed (Participants) | 70
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.2 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 40
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 70
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Subjects With Sustained Virologic Response (SVR12) 12 Weeks Post-treatment
Description: SVR12, defined as undetectable HCV RNA 12 weeks after the last day of study drug administration
Time Frame: 24 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Danoprevir,Ritonavir, Peg-IFN,RBV
Number analyzed (Participants) | 70
Participants | 66

ADVERSE EVENTS:
Arm/Group | Danoprevir,Ritonavir, Peg-IFN,RBV
Serious Adverse Events (participants affected / at risk) | 1/70
Other Adverse Events (participants affected / at risk) | 70/70
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danoprevir,Ritonavir, Peg-IFN,RBV (N=70)
acute pancreatitis (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Danoprevir,Ritonavir, Peg-IFN,RBV (N=70)
Neutrophil count decreased (Investigations) | 63 (85)
White blood cell decreased (Investigations) | 58 (69)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Ascletis, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

The study has been completed at all study sites for at least 3 years.